CLINICAL TRIAL: NCT06630559
Title: A Randomized, Active-Controlled, Double-Blind, Phase 3 Study to Compare Efficacy and Safety of CT-P55 with Cosentyx in Patients with Moderate to Severe Plaque Psoriasis
Brief Title: A Study to Compare Efficacy and Safety of CT-P55 and Cosentyx in Patients with Moderate to Severe Psoriasis
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-P55 3.1; 2024-513348-27 (EudraCT Number)
Record Dates: First submitted 2024-10-07; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- CT-P55 (Experimental)
  Interventions: Biological: CT-P55
- EU-approved Cosentyx (Active Comparator)
  Interventions: Biological: CT-P55; Biological: EU-approved Cosentyx

INTERVENTIONS:
Biological: CT-P55 — CT-P55, 300 mg by 2 subcutaneous (SC) injections of 150 mg/mL via Pre-Filled Syringe (PFS) every week for 5 doses (up to Week 4 after starting dose at Day 1), followed by every 4 weeks (Q4W) for 11doses (up to Week 48).
Biological: EU-approved Cosentyx — European Union (EU)-approved Cosentyx, 300 mg by 2 SC injections of 150 mg/mL via PFS every week for 5 doses (up to Week 4 after starting dose at Day 1), followed by Q4W for 11 doses (up to Week 48).
  Arms: EU-approved Cosentyx

SUMMARY:
The goal of this Phase 3 clinical trial is to compare efficacy and safety of CT-P55 with Cosentyx in patients with moderate to severe plaque psoriasis

DETAILED DESCRIPTION:
CT-P55 is a recombinant humanized monoclonal antibody containing the active ingredient secukinumab. CT-P55 is a drug product being developed by CELLTRION, Inc. and being compared to both the EU-approved Cosentyx®. In this study, Efficacy and Safety of CT-P55 will be evaluated in patients with Moderate to Severe Chronic Plaque Psoriasis.

ELIGIBILITY:
Inclusion Criteria:

- Patient has had a diagnosis of chronic plaque psoriasis for at least 24 weeks.

Exclusion Criteria:

* Patient diagnosed with forms of psoriasis other than chronic plaque-type or medication-induced psoriasis.
* Patient who has previously received Secukinumab or any other biologic drug directly targeting Interleukin-17 or the IL-17 receptor.
* Patient who has allergies to any of the excipients of study drug or materials of device or any other murine and human proteins, or patient with a hypersensitivity to immunoglobulin products.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Percent change from baseline in Psoriasis Area and Severity Index (PASI) score | Week 12

SECONDARY OUTCOMES:
Actual PASI scores | Up to 56 Weeks
Percent change from baseline in PASI score | Up to 56 Weeks
Proportion of patients who achieve at least 50/75/90/100% improvement from baseline in PASI (PASI 50/75/90/100) | Up to 56 Weeks
Proportion of patients with IGA score of clear (0) or almost clear (1) | Up to 56 Weeks
Change from baseline in Dermatology Life Quality Index (DLQI) | Up to 56 Weeks